CLINICAL TRIAL: NCT06891677
Title: COPD BALANCE: A Feasibility Study of Internet-Based Cognitive Behavioral Therapy and Educational Intervention to Improve Mental Health, Disease Knowledge, and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Internet-Based Cognitive Behavioral Therapy and Educational Program for People Living With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD BALANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonas Agholme (Other)
Responsible Party: Sponsor-Investigator, Jonas Agholme, Specialist in Internal Medicine, Department of Internal Medicine, Vrinnevi Hospital, Norrköping, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2024-06453-01
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Internet-based Cognitive Behavioral Therapy; Online CBT; Acceptance and Commitment Therapy; ACT; Educational intervention; Anxiety; Depression; Mental health; Quality of life; Feasibility study; Disease management; Pulmonary rehabilitation; Self-management education; Telehealth; Digital health; Respiratory medicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression; Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-group feasibility study in which all participants receive the same internet-based cognitive behavioral therapy (CBT) and educational intervention specifically designed for people with COPD. Outcomes will be assessed by comparing measures before and after the intervention on an individual level. Additionally, feasibility aspects such as recruitment rate, acceptability, adherence, and practicality of the intervention will be evaluated. No separate control group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Internet-Based CBT and Education for COPD (Experimental): Participants will receive an internet-based cognitive behavioral therapy (CBT) and educational program specifically designed for people with COPD. The intervention combines disease-specific education with CBT techniques, including elements of Acceptance and Commitment Therapy (ACT). The goal is to help participants manage COPD symptoms, reduce stress and anxiety, and improve their quality of life. Participants complete this 8-10-week online program at home.
  Interventions: Behavioral: Internet-Based Cognitive Behavioral Therapy (CBT) with ACT and COPD Education

INTERVENTIONS:
Behavioral: Internet-Based Cognitive Behavioral Therapy (CBT) with ACT and COPD Education — Participants receive an internet-based cognitive behavioral therapy (CBT) intervention combined with education specifically developed for COPD. The CBT program includes Acceptance and Commitment Therapy (ACT) components. The intervention lasts 8-10 weeks and consists of several online modules. Modules cover topics such as coping strategies, mindfulness techniques, disease knowledge, and symptom management. Participants complete the modules at home via a secure online platform, with regular support and feedback from trained healthcare professionals. The program aims to improve mental health, reduce anxiety and depression, enhance COPD knowledge, and help participants manage symptoms and daily life more effectively.
  Other Names: Internet-based CBT; Online CBT; Internet CBT; Acceptance and Commitment Therapy; Educational intervention for COPD

SUMMARY:
The goal of this clinical trial is to learn if an internet-based cognitive behavioral therapy (CBT) and education program can help improve mental health, disease knowledge, and quality of life in adults with chronic obstructive pulmonary disease (COPD). This is a feasibility study, meaning researchers want to find out if this online treatment program is practical, acceptable, and effective enough to use in a larger future study.

The main questions it aims to answer are:

Can internet-based CBT and disease education help participants feel less anxious, depressed, or stressed? Can this online program help participants better manage COPD symptoms and improve their quality of life? How easy and acceptable do participants find the online CBT and educational program?

Researchers will measure the following outcomes to see how well the program works:

Quantitative outcomes (using questionnaires and tests):

Depression symptoms (using Patient Health Questionnaire-9, PHQ-9) Anxiety symptoms (using Generalized Anxiety Disorder-7, GAD-7) Stress levels (using Perceived Stress Scale, PSS) Quality of life related to COPD (using St. George's Respiratory Questionnaire, SGRQ, and EuroQol-5 Dimensions, EQ5D) COPD-specific symptoms and impact on daily life (using COPD Assessment Test, CAT) Breathlessness severity during daily activities (using Modified Medical Research Council Dyspnea Scale, MRC) Physical capacity (using a 6-minute walk test) Lung function (using spirometry, a breathing test)

Qualitative outcomes (using interviews):

Participants' experiences and satisfaction with the internet-based therapy and education What participants think helps or hinders them from engaging with the online program How the program affects participants' daily lives and how they cope with COPD

Participants in the study will:

Take part in an internet-based CBT and education program designed specifically for COPD lasting 8-10 weeks. They can complete the program from home.

Answer questionnaires about mental health, stress, quality of life, COPD symptoms, and breathlessness before and after completing the program.

Visit the clinic two times (before and after the program) for breathing tests (spirometry) and physical capacity tests (6-minute walking test).

Some participants (10-15) will also participate in an interview to discuss their experiences and how they feel about the online treatment program.

The results of this study will help researchers understand whether internet-based CBT and COPD education is helpful and practical enough to study in a larger clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD).
* Access to a computer and stable internet connection.

Exclusion Criteria:

* Significant psychiatric illness requiring specialist psychiatric treatment by healthcare services within the last five years.
* Life expectancy less than six months.
* Dementia or cognitive impairment affecting the ability to participate.
* Limited proficiency in the Swedish language.
* Disabilities preventing computer use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Internet-Based CBT and Educational Intervention for COPD | At completion of the intervention (8-10 weeks)
  Feasibility is measured by participant adherence (how many complete at least 75% of the online program), acceptability (participant satisfaction through questionnaires and interviews), and recruitment rate (how quickly participants join the study). High feasibility means that participants find the intervention practical, acceptable, and manageable, indicating it could be used in a larger clinical trial.

SECONDARY OUTCOMES:
Change from Baseline in Depression Symptoms Measured by Patient Health Questionnaire-9 (PHQ-9) | Baseline (before intervention) and immediately after completing the intervention (8-10 weeks)
  Participants' symptoms of depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). This is a 9-item questionnaire that measures depression severity, with scores ranging from 0 (no depression) to 27 (severe depression). Researchers will assess if depression symptoms decrease after participants complete the internet-based CBT and educational intervention.
Change in Anxiety Symptoms Measured by Generalized Anxiety Disorder-7 (GAD-7) | Baseline and after completing the intervention (8-10 weeks)
  Anxiety is measured with the Generalized Anxiety Disorder-7 questionnaire, scoring from 0 (no anxiety) to 21 (severe anxiety). Lower scores after intervention indicate improvement.
Change in COPD-Related Quality of Life measured by St. George's Respiratory Questionnaire (SGRQ) | Baseline and immediately after completing the intervention (8-10 weeks)
  COPD-specific quality of life is measured using the St. George's Respiratory Questionnaire (SGRQ). Scores range from 0 to 100, with lower scores meaning better quality of life and fewer COPD symptoms.
Change in Health-Related Quality of Life Measured by EuroQol-5 Dimensions (EQ5D) | Baseline and after the intervention (8-10 weeks)
  General quality of life is measured with EuroQol-5 Dimensions (EQ5D). The EQ5D evaluates general health status across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate better quality of life.
Change in COPD Symptoms and Impact on Daily Life (COPD Assessment Test, CAT) | Baseline and after intervention completion (8-10 weeks)
  COPD symptoms and their impact on daily activities are measured using the COPD Assessment Test (CAT). Scores range from 0 to 40, where lower scores mean fewer COPD-related symptoms and problems.
Change in Breathlessness Severity (Modified Medical Research Council Dyspnea Scale, MRC) | Baseline and immediately after completing the intervention (8-10 weeks)
  Breathlessness during everyday activities is measured with the Modified Medical Research Council Dyspnea Scale (MRC). Scores range from 0 (breathless only during heavy exertion) to 4 (too breathless to leave the house). Lower scores after the intervention indicate improvement.
Change in Perceived Stress (Perceived Stress Scale, PSS-10) | Baseline and after completing the intervention (8-10 weeks)
  Stress levels are measured using the Perceived Stress Scale (PSS-10), with scores ranging from 0 (no stress) to 40 (high stress). The goal is to see if the intervention reduces participants' perceived stress.
Change in Physical Capacity (6-Minute Walk Test) | Baseline and after intervention (8-10 weeks)
  Physical capacity is measured with a 6-minute walk test (6MWT). Researchers measure how far participants can walk in six minutes, in meters, before and after the intervention to see if participants' physical ability improves.
Change in Lung Function (Spirometry, FEV1 and FVC) | Baseline and immediately after completing the intervention (8-10 weeks)
  Lung function is measured using spirometry, testing forced expiratory volume in one second (FEV1) and forced vital capacity (FVC).

OTHER OUTCOMES:
Participant Experiences of the Online Intervention (Qualitative Interviews) | At completion of intervention (8-10 weeks)
  Participants' experiences, satisfaction, and perceived impact of the online intervention are assessed through qualitative interviews. Researchers aim to understand participant views about barriers, benefits, and the intervention's impact on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Agholme, Medical Doctor, Principal Investigator — Region Östergötland
Locations (1):
- Lung- och allergimottagningen, Vrinnevisjukhuset, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to privacy considerations and ethical restrictions. Sharing individual participant data could risk compromising participant confidentiality and privacy.